CLINICAL TRIAL: NCT01843361
Title: Prevalence of Low Response to Clopidogrel in Patients After Acute Ischemic Stroke.
Brief Title: Clopidogrel Response in Acute Ischemic Stroke. The Bochumer CRISP Study
Acronym: Bo-CRISP
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Saskia Meves, MD, Ruhr University of Bochum
Other Study IDs: Meves-clopi-01
Record Dates: First submitted 2013-04-26; First posted 2013-04-30 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Ischemic Stroke
Keywords: Stroke; Clopidogrel; Aggregometry; Antiplatelet therapy; Platelet function tests
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- acute ischemic stroke: Determing cardiovascular risk factors or medication on clopidogrel response rates after an acute ischemic stroke

SUMMARY:
The aim of this study was to determine the prevalence rate and risk factors for chemical laboratory clopidogrel low-response (CLR) in the acute phase after an ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* acute ischemic stroke
* admittance to stroke unit
* clopidogrel medication

Exclusion Criteria:

* no consent
* prior bleeding disorders
* severe liver disorders
* current gastrointestinal disorders
* congestive heart failure
* life-threatening malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an acute ischemic stroke admitted to our stroke unit and treated with clopidogrel
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2010-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Result of platelet function test | one day
  Aggregometry result of antiplatelet therapy

CONTACTS AND LOCATIONS:
Overall Officials: Saskia H Meves, MD, Principal Investigator — Ruhr University Bochum, Department of Neurology
Locations (1):
- Department of Neurology, Ruhr University Bochum, Bochum, Germany

REFERENCES:
- [Background] Meves SH, Overbeck U, Endres HG, Krogias C, Neubauer H. Dose-dependent effect of early antiplatelet therapy in acute ischaemic stroke. Thromb Haemost. 2012 Jan;107(1):69-79. doi: 10.1160/TH11-06-0436. Epub 2011 Dec 8. PMID 22159509
- [Background] Fong J, Cheng-Ching E, Hussain MS, Katzan I, Gupta R. Predictors of biochemical aspirin and clopidogrel resistance in patients with ischemic stroke. J Stroke Cerebrovasc Dis. 2011 May-Jun;20(3):227-30. doi: 10.1016/j.jstrokecerebrovasdis.2009.12.004. Epub 2010 Jul 10. PMID 20621513